CLINICAL TRIAL: NCT00532623
Title: A Phase II Study of Gemcitabine in Combination With Vinorelbine vs. Sequential Gemcitabine Followed by Vinorelbine in Metastatic Breast Cancer
Brief Title: Phase II Study of Gemcitabine/Vinorelbine vs Sequential Gemcitabine Followed by Vinorelbine in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Jungsil Ro/MD, PhD, National Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-04-092
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2007-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination (Active Comparator)
  Interventions: Drug: Gemcitabine plus Vinorelbine
- Seqeuntial (Active Comparator): Gemcitabine monotherapy followed by Vinorelbine monotherapy:
  -Gemcitabine: 1,200 mg/m2, intravenously, on day 1 and day 8 in 3 week cycles. Vinorelbine: 30 mg/ m2, intravenously, on day 1 and day 8 in 3 week cycles.
  Interventions: Drug: Sequential

INTERVENTIONS:
Drug: Gemcitabine plus Vinorelbine — Gemcitabine, 1,000mg/m2 and Vinorelbine, 25mg/m2, on day 1 and day 8, every 3 week cycles
  Other Names: Gemzar; Navelbine
  Arms: Combination
Drug: Sequential — Gemcitabine monotherapy followed by Vinorelbine monotherapy:
  -Gemcitabine: 1,200 mg/m2, intravenously, on day 1 and day 8 in 3 week cycles. Vinorelbine: 30 mg/ m2, intravenously, on day 1 and day 8 in 3 week cycles.
  Other Names: Gemzar; Navelbine
  Arms: Seqeuntial

SUMMARY:
To evaluate the overall response rate of gemcitabine and vinorelbine combination (GV) and gemcitabine followed by vinorelbine (G⇒V) when used as palliative therapy in patients with stage IV and recurrent breast cancer.

DETAILED DESCRIPTION:
This is an open-label, randomized, two-arm, parallel group phase II study. Eligible patients will be randomized to each of the two treatment regimens, one of which is gemcitabine and vinorelbine combination therapy (Group A) and the other is gemcitabine monotherapy followed by vinorelbine monotherapy (Group B). Patients In group A monotherapy will receive gemcitabine and vinorelbine in combination, while patients in group B will receive gemcitabine monotherapy until the evidence of disease progression followed by vinorelbine. A total of 82 patients will be enrolled in this study. Patients will be randomized after stratified according to the number of prior chemotherapy including adjuvant chemotherapy and visceral disease. No maximum number of cycles is pre-determined. Patients may continue on study therapy until documented treatment failure.

Patients in group A who discontinue study therapy will proceed to the post-therapy follow-up phase of the study. Patients in group B who discontinue study therapy while treated with gemcitabine will proceed to receive vinorelbine on disease progression. Patients on vinorelbine who discontinue study therapy will proceed to the post-therapy follow-up phase of the study. Further treatment upon discontinuation of study therapy is at the discretion of the investigator.

A two arm, open label phase II study without control is appropriate for exploring the efficacy of gemcitabine with concurrent or sequential vinorelbine in this patient population and for evaluating and characterizing toxicities of two treatment approaches, qualitatively and quantitatively. The purpose of randomization in this phase II study is to diminish the possible impact of selection bias on treatment outcome and thus on interpretation of efficacy and safety data.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of stage IV or recurrent breast cancer.
* Previous anthracycline and/or taxane and/or capecitabine chemotherapy in adjuvant and metastatic setting.
* Previous hormonal therapy in adjuvant and metastatic setting.
* Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease.
* No other forms of cancer therapy, such as radiation, immunotherapy for at least 3 weeks before the enrollment in study.
* Performance status of 0, 1, 2 on the ECOG criteria.
* Clinically measurable disease, defined as unidimensionally measurable lesions with clearly defined margins on x-ray, CT scan, MRI or physical examination. Lesions serving as measurable disease must be at least 1cm by 1cm, as defined by x-ray, CT scan, MRI,or physical examination.
* Estimated life expectancy of at least 12 weeks.
* Patient compliance that allow adequate follow-up.
* Adequate hematologic (WBC count3,000/mm3, platelet count100,000/mm3), hepatic (bilirubin level1.5 mg/dL, AST, ALT3xULN), and renal (creatinine concentration 1.5 mg/dL) function.
* Informed consent from patient or patient's relative.
* Females at least 18 years of age.
* Childbearing women should use non-hormonal contraceptive method.

Exclusion Criteria:

* Previous chemotherapy > 3 for recurrent or stage IV disease Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence).
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-05; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
overall response rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, MD, PhD, Principal Investigator — National Cancer Center, Korea